CLINICAL TRIAL: NCT01462513
Title: LICC: L-BLP25 in Patients With Colorectal Carcinoma After Curative Resection of Hepatic Metastases - a Randomized, Placebo-controlled, Multicenter, Multinational, Double Blinded Phase II Trial
Brief Title: L-BLP25 in Patients With Colorectal Carcinoma After Curative Resection of Hepatic Metastases
Acronym: LICC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prof. Dr. Carl Schimanski (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Carl Schimanski, Coordinating Investigator, Johannes Gutenberg University Mainz
Organization: Johannes Gutenberg University Mainz (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LICC01
Record Dates: First submitted 2011-10-27; First posted 2011-10-31 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Colon Carcinoma; Rectum Carcinoma
Keywords: Colon carcinoma; Rectum carcinoma; Liver metastases
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — L-BLP25; MUC-1 monoclonal antibody

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L-BLP25 (Experimental): L-BLP25 treatment
  Interventions: Biological: L-BLP25
- Placebo (Placebo Comparator): Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: L-BLP25 — Treatment: 930µg per treatment once weekly for 8 weeks, then at 6-week intervals during years 1 and 2.
  Other Names: MUC1-antibody
  Arms: L-BLP25
Biological: Placebo — Treatment: Placebo 930µg per treatment, once weekly for 8 weeks, then at 6-week intervals during years 1 and 2.
  Arms: Placebo

SUMMARY:
Comparative evaluation of recurrence-free survival (RFS) time and 3 year overall survival (OS) time between the treatment groups (L-BLP25 plus cyclophosphamide versus placebo and saline infusion).

DETAILED DESCRIPTION:
This trial is designed for patients with metastatic colorectal carcinoma (CRC), who have undergone a complete resection of their primary tumor and recent resection of their liver metastases (R0 or R1) with curative intent. No generally accepted standard care is available following curative-intent resection of hepatic metastases in colorectal cancer patients. L-BLP25 is a cancer vaccine that targets MUC1, a well known tumor-associated antigen. Recently, it has been shown that MUC1 is associated with cellular transformation as demonstrated by tumorigenicity and can confer resistance to genotoxic agents. High levels of MUC1 cell surface expression, reported immunosuppressive activities of its released ectodomain, and anti-adhesive properties all contribute to the ability of the MUC1 antigen to protect and promote tumor cell growth and survival, and make MUC1 an attractive target for cancer immunotherapy.

Based on these results, L BLP25 may have potential as adjuvant therapy after curative resection of hepatic metastases in colorectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Female patients of childbearing potential (and if appropriate male patients with female partners of childbearing potential) must be willing to use an adequate method of contraception for 4 weeks prior to, during and 12 weeks after the last dose of trial medication. A negative pregnancy test is required for female subjects. Adequate contraception for female subjects is defined as two barrier methods, or one barrier method with a spermicide, or intrauterine device or use of hormonal female contraceptive.
* Histologically confirmed diagnosis of adenocarcinoma of the colon or rectum with complete resection of primary tumor and no evidence of local relapse.
* Metastatic disease of the liver, with recent (< 8 weeks prior to randomization), both primary or secondary resection (R0 or R1) of all liver metastases. Metastasectomy may have been either synchronous or metachronous. Neoadjuvant therapy may have been applied prior to metastasectomy.
* Subject has had a colonoscopy or rectoscopy within the last three months prior to initiation of therapy
* Subject has an ECOG performance status of 0 or 1.
* Subject has adequate hematologic, hepatic, and renal function within 2 weeks prior to initiation of therapy as defined by the following: Absolute neutrophils > 1,500/mm3 and platelets > 140,000/mm3. Bilirubin < 1.5 x upper limit of normal (ULN). AST and ALT < 2.5 x ULN. Creatinine < 1.5 x ULN.
* International Normalized Ratio (INR) and partial thromboplastin time (PTT) within normal range respectively within therapeutic range in case of anticoagulation.
* Willingness to comply with study protocol requirements.

Exclusion Criteria:

* Metastases other than liver metastases.
* R2 and Rx resected liver metastases. Patients with R1 resected liver metastases can be included if a further surgical resection is seen as not indicated or necessary in the surgeon´s opinion.
* Chemotherapy within 4 weeks prior to randomization.
* Receipt of immunotherapy (e.g. interferons, tumor necrosis factor, interleukins, or growth factors [GM-CSF, G-CSF, M- CSF], monoclonal antibodies) within 4 weeks (28 days) prior to randomization.
* Any known autoimmune disease, past or current.
* A recognized immunodeficiency disease including cellular immuno-deficiencies, hypogammaglobulinemia or dysgammaglobulinemia; hereditary or congenital immunodeficiencies.
* Known or newly diagnosed active hepatitis B infection and/or hepatitis C infection, autoimmune hepatitis, known human immunodeficiency virus infection, or any other infectious process that in the opinion of the investigator could compromise the subject's ability to mount an immune response, or expose him/ her to likelihood of more and/or severe side effects.
* Past or current history of malignant neoplasm other than CRC, except for curatively treated non-melanoma skin cancer, in-situ carcinoma of the cervix or other cancer curatively treated and with no evidence of disease for at least 5 years.
* Medical or psychiatric conditions that would interfere with ability to provide informed consent, communicate side effects, or comply with protocol requirements.
* Clinically significant cardiac disease, e.g. cardiac failure of New York Heart Association classes III-IV; uncontrolled angina pectoris, uncontrolled arrhythmia, uncontrolled hypertension, myocardial infarction in the previous 12 months as confirmed by an ECG.
* Splenectomy.
* Previous (less than 4 weeks prior to randomization) or concurrent treatment with a non-permitted drug.
* Pregnancy and lactation period.
* Participation in another clinical study within 30 days prior to randomization.
* Known hypersensitivity to the study treatment drugs.
* Known alcohol or drug abuse.
* Legal incapacity or limited legal capacity.
* Any other reason that, in the opinion of the investigator, precludes the subject from participating in this study.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2011-08; Primary Completion 2017-12-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Comparative evaluation of recurrence-free survival (RFS) time and 3 year overall survival (OS) time between the treatment groups (L-BLP25 plus cyclophosphamide versus placebo and saline infusion). | until December 2017
  The primary variable of this trial is recurrence free survival (RFS) time. RFS time will be measured from the date of randomization to the date of recurrence. For subjects not known to have experienced recurrence or death at the time of analysis, the time between the date of randomization and the date of last evaluation for recurrence will be calculated and used as a censored observation in the analysis.

SECONDARY OUTCOMES:
Safety / Tolerability | until December 2017
  Assessment of safety will include:
  * AEs, SAEs
  * Vital signs (body temperature, respiratory rate, heart rate, and blood pressure) and physical examinations,
  * Clinical laboratory assessments from hematology and biochemistry samples
Recurrence-free survival time in the subgroup of MUC1 positive cancers | until December 2017
  Recurrence free survival (RFS) time of MUC1 positive cancers will be measured from the date of randomization to the date of relapse based on standard imaging. For subjects not known to have experienced recurrence or death at the time of analysis, the time between the date of randomization and the date of last evaluation for recurrence or death will be calculated and used as a censored observation in the analysis.
Overall survival time in a subgroup of MUC1 positive cancers | until December 2017
  Overall survival time of MUC1 positive cancers will be measured from the date of randomization to the date of death. For subjects not known to be deceased at the time of analysis, the time between the date of randomization and the date of last contact, or date lost to follow-up, will be calculated and used as a censored observation in the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Carl Christoph Schimanski, Prof. Dr., Principal Investigator — Universitätsmedizin Mainz
Locations (21):
- Salzburger Universitätsklinikum, Universitätsklinik für Innere Medizin III, Salzburg, Austria
- Germany (20):
  - Klinikum Altenburger Land, Altenburg
  - Campus Virchow-Klinikum, Charite Centrum 8, Berlin
  - Klinikum Darmstadt, Darmstadt
  - Universitätsklinikum Essen WTZ-Ambulanz, Innere Medizin (Tumorforschung), Essen
  - Klinik für Allgemeine Innere Medizin, Onkologie / Hämatologie, Esslingen am Neckar
  - Klinikum der Johann W- Goethe Unversität, Klinik für Allgemein- und Viszeralchirurgie, Frankfurt
  - Onkologische Schwerpunktpraxis Eppendorf, Hamburg
  - Städtisches Klinikium Abt. Allgemein- und Visceralchirurgie, Karlsruhe
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum Magdeburg, Magdeburg
  - Universitätsmedizin Mainz, Mainz
  - Universtitäsmedizin Gießen und Marburg, Marburg
  - Praxis für Hämatologie und Onkologie, Mülheim
  - Klinikum der Universität München-Grosshadern, Medizinische Klinik III, München
  - GP für Hämatologie und Onkologie Offenburg, Offenburg
  - Oncologianova GmbH, Recklinghausen
  - Universitätsklinikum Regensburg, Regensburg
  - Robert-Bosch Krankenhaus, Zentrum für Innere Medizin, Stuttgart
  - Krankenhaus der Barmherzigen Brüder, Trier
  - Klinikum Weiden, Medizinische Klinik I, Weiden

REFERENCES:
- [Derived] Schimanski CC, Kasper S, Hegewisch-Becker S, Schroder J, Overkamp F, Kullmann F, Bechstein WO, Vohringer M, Ollinger R, Lordick F, Heinemann V, Geissler M, Schulz-Abelius A, Bernhard H, Schon MR, Greil R, Galle P, Lang H, Schmidtmann I, Moehler M. Adjuvant MUC vaccination with tecemotide after resection of colorectal liver metastases: a randomized, double-blind, placebo-controlled, multicenter AIO phase II trial (LICC). Oncoimmunology. 2020 Aug 23;9(1):1806680. doi: 10.1080/2162402X.2020.1806680. PMID 32923171